CLINICAL TRIAL: NCT06364683
Title: The Relationship Between Exercise Adherence, Self-Efficacy, and Health Literacy in Patients With Coronary Artery Disease: A Descriptive Correlational Study
Brief Title: Coronary Artery Disease and Exercise Adherence
Status: Completed | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Seyma Demir, Assistant Professor, Abant Izzet Baysal University
Other Study IDs: AIBU-HSF-SDEMIR-04
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Adherence, Treatment; Coronary Artery Disease
Keywords: exercise adherence; coronary artery disease; self-efficacy; health literacy
MeSH Terms: conditions — Treatment Adherence and Compliance; Coronary Artery Disease | interventions — Longitudinal Studies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey study — The data collection tools to be used in the study will be filled. It does not include any invasive or non-invasive intervention.

SUMMARY:
This study aims to determine the factors affecting exercise adherence in patients with coronary artery disease (CAD). For this purpose, the following measurement tools will be used respectively: (1) "Patient Information Form" including sociodemographic characteristics of the patients and medical information related to the disease, (2) the Exercise Adherence Rating Scale (EARS), (3) Exercise Self-Efficacy Scale (ESE) and, (4) Turkish-Health Literacy Survey Europe-Q12 (HLS-EU-19-12Q-TR). Statistical analyses will be carried out by descriptive statistics (number, percentage, mean, standard deviation, etc.), correlation analysis and regression analysis.

DETAILED DESCRIPTION:
Coronary Artery Disease (CAD) is the most common form of cardiovascular disease in the world and is one of the leading causes of mortality and morbidity in Turkey and worldwide. Exercise training is very important in the treatment of CAD because of its various cardiovascular benefits. However, most patients have been shown to have low to moderate adherence rates to the recommended exercise prescription. The results of a limited number of studies show that the factors affecting exercise adherence in patients with CAD need to be supported by new studies. This study aims to determine the factors affecting exercise adherence in patients with coronary artery disease (CAD). The study will be conducted with CAD patients followed up in the cardiology clinics of a tertiary care hospital in northern Turkey. A cohen's d will be calculated using preliminary data from 20 patients using Exercise Adherence Rating Scale (EARS), and an adequate sample size will be determined with a 95% confidence interval, a bias level of 0.05, and 80% power. Patients with a diagnosis of CAD confirmed by a physician at least one year ago, who have been recommended any exercise/physical activity by a physician according to article 1 of EARS, who are ≥18 years old and <75 years old, and who have the ability to understand and speak Turkish will be included in the study. The data will be collected using the following measurement tools respectively: (1) "Patient Information Form" including sociodemographic characteristics of the patients and medical information related to the disease, (2) the Exercise Adherence Rating Scale (EARS), (3) Exercise Self-Efficacy Scale (ESE) and, (4) Turkish-Health Literacy Survey Europe-Q12 (HLS-EU-19-12Q-TR). Statistical analyses will be carried out by descriptive statistics (number, percentage, mean, standard deviation, etc.), correlation analysis and regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of CAD confirmed by a physician at least one year ago,
* Individuals who have been recommended any exercise/physical activity by a physician according to item 1 of the EARS,
* Turkish comprehension and speaking skills.

Exclusion Criteria:

* Presence of serious physical and mental health problems,

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population refers to adults with coronary artery disease.
Sampling Method: Probability Sample
Enrollment: 208 (Actual)
Dates: Start 2024-05-13 (Actual); Primary Completion 2024-11-13 (Actual); Study Completion 2025-05-13 (Actual)

PRIMARY OUTCOMES:
exercise adherence | Baseline
  EARS, a self-report measurement tool, was developed to assess adherence to prescribed home exercise regimes. It has three sections, A (qualitative information about participants' exercise adherence behaviours), B (exercise adherence behaviours) and C (factors preventing and facilitating exercise). Sections B and C are scored using a 5-point Likert scale (0=totally agree to 4=totally disagree).The total scores of Parts B and C range from 0 to 24 and 0 to 40, respectively, and the possible total scores (Part B + Part C) range from 0 to 64. A higher total score from the EARS indicates better exercise adherence. Cronbach's alpha coefficient was found to be 0.81 in the original scale and 0.86 in the Turkish version.
predictors for exercise adherence | Baseline
  The following instruments will be used to measure predictors for exercise adherence: (1) patient information form, (2) ESE and, (3) HLS-EU-19-12Q-TR. The patient information form includes 14 items including sociodemographic characteristics and medical information related to the disease. The ESE has 18 items. Scores between 0-100% are obtained from the scale, the higher the score, the higher the self-efficacy level of the participants. Cronbach's alpha coefficient is 0.94. The HLS-EU-19-12Q-TR has 12 items. The total score is calculated with a standardised index score (Index=[mean-1]*[50/3]). The standardised index score varies between 0-50. A score of 33 and over indicates adequate literacy. Correlation analyses and regression modelling will be used for the factors affecting participants' exercise adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Şeyma Demir Erbaş, PhD, Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Şeyma Demir Erbaş, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Participant data will not be shared openly with other researchers due to the confidentiality of personal data. The primary investigator of the study can be contacted for data sharing.